CLINICAL TRIAL: NCT06763237
Title: Abdominal Transcutaneous Electrical Acupoint Stimulation on Children With Autism Spectrum Disorder: A Randomized Clinical Trial
Brief Title: Abdominal Transcutaneous Electrical Acupoint Stimulation on Children With Autism Spectrum Disorder
Acronym: TEAS/ASD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Xian Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJTU1AF2024LSYY-352; 82305315 (Other Grant/Funding Number: The National Natural Science Foundation of China)
Record Dates: First submitted 2024-11-18; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder; Autism in Children
Keywords: Transcutaneous electrical acupoint stimulation; Gastrointestinal symptoms; Children; Autism spectrum disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Interventional Study Model is consisted of ABA therapy combined with TEAS treatment or sham TEAS treatment. The common ABA therapy can be effective for anyone, including any child with ASD. Each specific rehabilitation training method of ABA has its own characteristics: DTT (Discrete TrialTraining) is critical to the establishment of attention, listening to commands and other abilities; VB (Verbal Behavior) is very helpful for language ability; PRT (Pivotal Response Treatment) has an obvious effect on children who are severely affected; NET (Natural Education Training)helps to generalize the content in one-to-one courses. Following randomization, participants had an appointment with the TEAS operator. The Zhongwan (RN 12), bilateral Tianshu (ST 25), Qihai (RN 6) and Guanyuan (RN 4) acupoints were selected according to the concept of traditional Chinese medicine that specialized in treating gastrointestinal diseases, improving intestinal function.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABA Therapy with active TEAS (Active Comparator): The TEAS intervention is delivered using an electroacupuncture device (SDZ-V, Hwato, Soochow Medical Instruments Co., Ltd., China). Self-adhesive electrodes are placed at acupoints Zhongwan (RN12), bilateral Tianshu (ST25), Qihai (RN6), and Guanyuan (RN4). Stimulation is applied using dense-sparse wave alternating frequencies (3 Hz for 2 s cycles) at an intensity of 3-10 mA, adjusted to the participant's tolerance. Each session lasts 30 minutes, conducts once daily, five days per week, for a total of 40 sessions.
  The ABA therapy focuses on enhancing skills in areas such as social interaction, communication, academics, motor function, and self-care. Each session lasts 30 minutes, conducts once daily, five days per week, for a total of 40 sessions.
  Interventions: Device: abdominal transcutaneous electrical acupoint stimulation (abdominal TEAS)
- ABA Therapy with Sham TEAS (Sham Comparator): The sham TEAS intervention is delivered using an electroacupuncture device (SDZ-V, Hwato, Soochow Medical Instruments Co., Ltd., China). Self-adhesive electrodes are placed at acupoints Zhongwan (RN12), bilateral Tianshu (ST25), Qihai (RN6), and Guanyuan (RN4). Stimulation is applied using dense-sparse wave alternating frequencies (3 Hz for 2 s cycles) at an intensity of 0 mA. Each session lasts 30 minutes, conducts once daily, five days per week, for a total of 40 sessions.
  ABA therapy focuses on enhancing skills in areas such as social interaction, communication, academics, motor function, and self-care. Each session lasts 30 minutes, conducts once daily, five days per week, for a total of 40 sessions.
  Interventions: Device: abdominal transcutaneous electrical acupoint stimulation (abdominal TEAS)

INTERVENTIONS:
Device: abdominal transcutaneous electrical acupoint stimulation (abdominal TEAS) — The TEAS intervention is delivered using an electroacupuncture device (SDZ-V, Hwato, Soochow Medical Instruments Co., Ltd., China). Self-adhesive electrodes are placed at acupoints Zhongwan (RN12), bilateral Tianshu (ST25), Qihai (RN6), and Guanyuan (RN4). Stimulation is applied using dense-sparse wave alternating frequencies (3 Hz for 2 s cycles) at an intensity of 3-10 mA, adjusted to the participant's tolerance. Each session lasts 30 minutes, conducts once daily, five days per week, for a total of 40 sessions.
  The ABA therapy focuses on enhancing skills in areas such as social interaction, communication, academics, motor function, and self-care. ABA is delivered in a variety of settings, including school, home, clinic, and other community settings. The goal of treatment is to help children function as independently and successfully as possible. Each session lasts 30 minutes, conducts once daily, five days per week, for a total of 40 sessions.
  Other Names: TEAS; Applied Behavior Analysis (ABA) therapy

SUMMARY:
The goal of this clinical trial is to learn if abdominal transcutaneous electrical acupoint stimulation (abdominal TEAS) works to treat autism spectrum disorder (ASD) in children. It will also learn about the safety of abdominal TEAS. The main questions it aims to answer are:

Does abdominal TEAS a safe and effective treatment for children with autism spectrum disorder and gastrointestinal symptoms? Researchers will compare abdominal TEAS to a placebo (a sham abdominal TEAS without stimulation) to see if abdominal TEAS works to treat ASD.

Participants will:

Take abdominal TEAS or sham abdominal TEAS 5 days a week for 8 weeks. Visit the clinic once every 4 weeks for checkups and tests Keep a diary of their symptoms.

DETAILED DESCRIPTION:
Following randomization, participants had an appointment with the TEAS operator. The TEAS operators had a minimum of 2 years of experience in acupuncture treatment and held a membership with a national professional association in China. The Zhongwan (RN 12), bilateral Tianshu (ST 25), Qihai (RN 6) and Guanyuan (RN 4) acupuncture points were selected according to the concept of traditional Chinese medicine that specialized in treating gastrointestinal diseases, improving intestinal function, and eliminating various symptoms caused by intestinal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed as autism based on the DSM-V and Autism Diagnostic Observation Schedule, Second Edition (ADOS-2)
* Aged 3 to 6 years

Exclusion Criteria:

* Diagnosed with other organic diseases (such as severe hearing and visual impairment, brain trauma) and neurological disease (e.g., epilepsy, Rett syndrome), or psychiatric disorder (schizophrenia, bipolar affective disorder, etc)
* Oral or injected antibiotics within 30 days before screening
* History of acupuncture, electroacupuncture, TEAS treatment before screening
* Taking antipsychotic drugs and psychobiotic supplements within 30 days before screening

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale (CARS) | From enrollment to the end of treatment at 8 weeks, and follow up to 16 weeks.
  CARS is a 15 item behavioral rating scale developed to identify children with autism and to categorize these behaviors from mild to moderate to severe.

SECONDARY OUTCOMES:
The Clinical Global lmpression - lmprovement scale (CGI-I) | From enrollment to the end of treatment at 8 weeks, and follow up to 16 weeks.
  The Clinical Global Impression Scale (CGI) is a 7-point scale that has been adapted so that clinicians can easily and quickly rate social communication behaviors.
Social Responsiveness Scale-2 (SRS-2) | From enrollment to the end of treatment at 8 weeks, and follow up to 16 weeks.
  The Social Responsiveness Scale-2 (SRS-2) measures the presence and severity of social impairments within the autism spectrum. Parents, teachers, or other observers evaluate social abilities in various natural settings for children between 2.5 and 18 years using age-appropriate forms with 65 Likert-scale items. SRS-2 has 5 subscales: social awareness, social cognition, social communication, social motivation, restricted interests, and repetitive behavior. The total continuous score indicates the severity of social deficits in the autism spectrum.
Autism Treatment Evaluation Checklist (ATEC) | From enrollment to the end of treatment at 8 weeks, and follow up to 16 weeks.
  The Autism Treatment Evaluation Checklist (ATEC) is a method to assess how an individual with autism is progressing over time. It was developed with the aim of evaluating a wide array of behaviors and skills, thereby offering a comprehensive look at an individual's abilities and challenges. This makes it a valuable tool for tracking the effectiveness of various autism treatments. It is designed to be filled out by individuals who know the person with autism well, such as parents or primary caregivers, and can be completed in approximately 10-20 minutes. The ATEC spans four subtests: Speech/Language/Communication、Sociability、Sensory/Cognitive Awareness、Health/Physical/Behavior. These subtests evaluate various aspects, including verbal and non-verbal communication skills, social interactions, sensory responses, cognitive abilities, physical health, and behaviors.
Gastrointestinal Symptom Rating Scale (GSRS) | From enrollment to the end of treatment at 8 weeks, and follow up to 16 weeks.
  The GSRS is self-administered scale and has 15 questions divided into 5 domains that cover the gastrointestinal system: diarrhea, constipation, abdominal pain, reflux and indigestion. The scale answers are arranged according to the 4-point Likert scale, in which "1" indicates absence and "4" the higher frequency or intensity of the symptoms. This tool has already been validated as to their questions and assessment scales (construct validity and criterion validity).
6-Item Gastrointestinal Severity Index (6-GSI) | From enrollment to the end of treatment at 8 weeks, and follow up to 16 weeks.
  The severity of GI symptoms was assessed using a shortened version of the 6-item Gastrointestinal Severity Index (6-GSI) questionnaire, composed of six symptoms, including constipation, diarrhea, stool consistency, stool smell, flatulence, and abdominal pain. Each symptom is rated on a three-point Likert-type scale ranging from 0 to 2, with a higher score signifying more severe GI symptoms.
Bristol Stool Scale (BSS) | From enrollment to the end of treatment at 8 weeks, and follow up to 16 weeks.
  The Bristol Stool Scale (BSS) is a 7-point scale used extensively in clinical practice and research for stool form measurement. This is a tool to assist patients, family members and health care providers to share common language about stool consistency. The original Bristol Stool Form Scale description with notations in brackets: Type 1 Separate hard lumps, like nuts [constipation/encopresis, difficult to pass] Type 2 Sausage-shaped but lumpy Type 3 Like a sausage or snake but with cracks on its surface Type 4 Like a sausage or snake, smooth and soft [average stool] Type 5 Soft blobs with clear-cut edges Type 6 Fluffy pieces with ragged edges, a mushy stool Type 7 Watery, no solid pieces. [diarrhea, easy to pass and may involuntarily be passed]
Differences in gut microbiota composition | From enrollment to the end of treatment at 8 weeks.
  Differences in gut microbiota composition in children with ASD before and after intervention. It involves studying the collective genomes of microorganisms that reside in the gastrointestinal tract. This approach aims to understand the composition, diversity, and functional potential of the microbiota, which plays a crucial role in human health and well-being. By analyzing the DNA extracted directly from fecal samples, researchers can identify and characterize the various bacterial, viral, and fungal species present in the gut.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The first affiliated hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xi'an Children's Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Yes
Baseline characteristics of patients, the primary and secondary outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Ending 2 years after the publication of results.
Access Criteria: The IPD is available for sharing with qualified researchers or organizations upon request. The researchers must meet to be eligible for accessing IPD, such as having a scientifically sound research proposal, being affiliated with an academic institution or research organization, and having appropriate ethical approval. Researchers must agree to a data use agreement that outlines the terms and conditions of using the shared IPD, including confidentiality, data security, and intellectual property rights. The registry should submit a research proposal, reviewing the proposal by an independent committee, and granting access once the proposal is approved. The shared IPD is protected from unauthorized access, use, or disclosure, and that appropriate measures are in place to maintain participant confidentiality and privacy. The researchers can access IPD by contact the principle investigator of this study.

REFERENCES:
- [Result] Zhuo L, Zhao X, Zhai Y, Zhao B, Tian L, Zhang Y, Wang X, Zhang T, Gan X, Yang C, Wang W, Gao W, Wang Q, Rohde LA, Zhang J, Li Y. Transcutaneous electrical acupoint stimulation for children with attention-deficit/hyperactivity disorder: a randomized clinical trial. Transl Psychiatry. 2022 Apr 21;12(1):165. doi: 10.1038/s41398-022-01914-0. PMID 35449191
- [Result] Adams JB, Johansen LJ, Powell LD, Quig D, Rubin RA. Gastrointestinal flora and gastrointestinal status in children with autism--comparisons to typical children and correlation with autism severity. BMC Gastroenterol. 2011 Mar 16;11:22. doi: 10.1186/1471-230X-11-22. PMID 21410934
- [Result] Toolan C, Holbrook A, Schlink A, Shire S, Brady N, Kasari C. Using the Clinical Global Impression scale to assess social communication change in minimally verbal children with autism spectrum disorder. Autism Res. 2022 Feb;15(2):284-295. doi: 10.1002/aur.2638. Epub 2021 Nov 19. PMID 34800004
- [Result] Mensi MM, Rogantini C, Marchesi M, Borgatti R, Chiappedi M. Lactobacillus plantarum PS128 and Other Probiotics in Children and Adolescents with Autism Spectrum Disorder: A Real-World Experience. Nutrients. 2021 Jun 14;13(6):2036. doi: 10.3390/nu13062036. PMID 34198499
- [Result] Dai Y, Zhang L, Yu J, Zhou X, He H, Ji Y, Wang K, Du X, Liu X, Tang Y, Deng S, Langley C, Li WG, Zhang J, Feng J, Sahakian BJ, Luo Q, Li F. Improved symptoms following bumetanide treatment in children aged 3-6 years with autism spectrum disorder: a randomized, double-blind, placebo-controlled trial. Sci Bull (Beijing). 2021 Aug 15;66(15):1591-1598. doi: 10.1016/j.scib.2021.01.008. Epub 2021 Jan 16. PMID 36654288
- [Result] Hirota T, King BH. Autism Spectrum Disorder: A Review. JAMA. 2023 Jan 10;329(2):157-168. doi: 10.1001/jama.2022.23661. PMID 36625807
- See also: Related Info — https://www.medicalresearch.org.cn/clinicalResearch/researchInfo?id=67587e4d-2bf5-4cda-88c2-cf10fea5b21a